CLINICAL TRIAL: NCT04894331
Title: Diet Intervention Study Through Telemedicine Assistance on SNAS Patients in COVID-19 Pandemic
Brief Title: Telemedicine for SNAS Patients in COVID-19 Pandemic
Acronym: DISTANCE
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Eleonora Nucera, Head of Allergy Unit, Catholic University of the Sacred Heart
Other Study IDs: ID 3448
Record Dates: First submitted 2021-05-18; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Systemic Nickel Allergic Syndrome
Keywords: Food Allergy; COVID-19; Telemedicine; Telenutrition; Quality of Life; Systemic Nickel Allergic Syndrome
MeSH Terms: conditions — Food Hypersensitivity; COVID-19 | interventions — Diet Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SNAS patients: Patients with (a) history of SNAS (coexistence of typical cutaneous and gastrointestinal symptoms); (b) positive Ni-patch test; (c) clinical improvement of at least 70% from baseline after 4 weeks of low-Ni diet; (d) positivity of a double-blind placebo-controlled oral Ni challenge (DBPCO). Exclusion criteria include (a) age < 18 years and >65 years; (b) other organic gastrointestinal diseases, such as peptic ulcer, inflammatory bowel diseases, celiac disease, gastrointestinal infections, and small intestinal bacterial overgrowth; (c) diabetes mellitus; (d) hepatic, renal or cardiac dysfunction; (e) thyroid disease or tumour; (f) concomitant treatment with steroids and/or antihistamines in the previous 4 weeks; (g) pregnancy and lactation; (h) smoking, abuse of alcohol, coffee, tea, and cola intake, and (i) inability to give written informed consent.
  Interventions: Other: Dietary intervention; Other: Video call

INTERVENTIONS:
Other: Dietary intervention — Each patient receives one of 5 dietary plans, different only for energy intake (1400-1600-1800-2000-2100 Kcal/day). The choice depends on the personalized energy needs. The energy requirement is calculated on basal metabolic rate (BMR) of the patient according to Harris & Benedict's and Schofield's formulas.
  All dietary plans include foods with low-Ni content. Finally, each patient completes 30-day personalized diet.
  Other Names: Diet therapy
Other: Video call — Each patient receives a follow-up remote visit through video call 15 and 30 days after the start of the dietary intervention.
  Other Names: Telenutrition tool

SUMMARY:
Restrictions due to Covid-19 pandemic have brought negative social and psychological consequences on people and limited patients' access to hospital care.

In this context, "telemedicine" and, specifically, "tele-nutrition" (in nutritional field) allows remotely monitor and support food allergic patients subjected to restricted diets using information and communication technologies.

The investigators focus attention on patients with diagnosis of Systemic Nickel Allergic Syndrome (SNAS) undergoing low-nickel diet to evaluate nutritional and psychological states through tele-nutrition tools during COVID-19 pandemic.

The aims of this study are: (a) to investigate dietary-nutritional status and, (b) to assess quality of life and adherence to dietary therapy before and after 30-day personalized diet therapy through tele-nutrition tools.

Each subject enrolled in the study goes allergological work-up to assess diagnosis of SNAS and following procedures: (a) face-to-face visit (nutritional visit and quality of life evaluation) concluding with prescription of one of five personalized and balanced dietary plans different for calory intake, (b) video call visit for dietary evaluation and assessment of adherence to diet after 15 days, and (c) video call visit for dietary and quality of life evaluation and assessment of adherence to diet therapy after 30 days (end of study).

DETAILED DESCRIPTION:
There are no previous studies focused on the tele-nutrition for the evaluation of dietary-nutritional status of patients suffered from Systemic Nickel Allergic Syndrome (SNAS).

The aims of this study are (a) to investigate dietary-nutritional status (primary outcome) and, (b) to assess quality of life (QoL) and adherence to dietary therapy (secondary outcomes) of SNAS patients before and after personalized diet therapy through tele-nutrition tools at time of COVID-19 pandemic.

The investigators perform a prospective, single-center, observational study enrolling SNAS patients in order to evaluate dietary-nutritional status and QoL, before and after 30-day personalized diet therapy, and adherence to low Ni diet, through tele-nutrition tools, during COVID-19 pandemic.

The study is performed at the Allergology Unit and Dietetics and Clinical Nutrition Unit of Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome, Italy.

All enrolled patients give their signed informed consent to participation in the study.

The investigators enroll patients with (a) history of SNAS (coexistence of typical cutaneous and gastrointestinal symptoms); (b) positive Nickel (Ni)-patch test; (c) clinical improvement of at least 70% from baseline after 4 weeks of low-Ni diet; (d) positivity of a double-blind placebo-controlled oral Ni challenge (DBPCO). Exclusion criteria include (a) age < 18 years and >65 years; (b) other organic gastrointestinal diseases, such as peptic ulcer, inflammatory bowel diseases, celiac disease, gastrointestinal infections, and small intestinal bacterial overgrowth; (c) diabetes mellitus; (d) hepatic, renal or cardiac dysfunction; (e) thyroid disease or tumour; (f) concomitant treatment with steroids and/or antihistamines in the previous 4 weeks; (g) pregnancy and lactation; (h) smoking, abuse of alcohol, coffee, tea, and cola intake, and (i) inability to give written informed consent.

Patients go pre-diet face-to-face visit (time 0, T0), complete 30-day personalized diet and, then, go follow-up remote visit through video call (time 2, T2). A further video call is performed 15 days after the start of the diet therapy treatment (time 1, T1).

The study uses the commercially available online platform Microsoft Teams, which is included in the Fondazione Policlinico Universitario A. Gemelli IRCCS's Microsoft Office 365 package.

Variables The investigators select two primary outcome measurements (dietary assessment and anthropometric data) to evaluate dietary-nutritional status of SNAS patients. Moreover, the investigators adopt Short-Form 36-Item Health Survey (SF-36v2) questionnaire as tool to evaluate QoL (secondary outcome). Finally, adherence to diet therapy (secondary outcome) is investigated through video call at T1 and T2.

Measurement

Study procedures:

T0 face-to-face visit:

* Dietary assessment: nutritional history and eating habits.
* Collection of anthropometric data.
* QoL evaluation. Each patient answers SF-36v2 (Italian version) questionnaire. At the end of visit, each patient receives one of 5 dietary plans, different only for energy intake (1400-1600-1800-2000-2100 Kcal/day). The choice depended on the personalized energy needs.

All dietary plans include foods with low-Ni content.

T1 video call visit:

* Dietary assessment: collection of anthropometric data.
* Assessment of adherence to dietary therapy through question "How many days a week did the participant adhere to the prescribed dietary treatment? - Two possible mutually exclusive answers: 1) <5 days a week, 2) ≥ 5 days a week.

T2 video call visit:

* Dietary evaluation: collection of anthropometric data.
* Assessment of adherence to the dietary treatment.
* QoL evaluation.

ELIGIBILITY:
Inclusion Criteria:

* history of SNAS (coexistence of typical cutaneous and gastrointestinal symptoms);
* positive Ni-patch test;
* clinical improvement of at least 70% from baseline after 4 weeks of low-Ni diet;
* positivity of a double-blind placebo-controlled oral Ni challenge (DBPCO).

Exclusion Criteria:

* age < 18 years and >65 years;
* other organic gastrointestinal diseases, such as peptic ulcer, inflammatory bowel diseases, celiac disease, gastrointestinal infections, and small intestinal bacterial overgrowth;
* diabetes mellitus;
* hepatic, renal or cardiac dysfunction;
* thyroid disease or tumour;
* concomitant treatment with steroids and/or antihistamines in the previous 4 weeks;
* pregnancy and lactation;
* smoking, abuse of alcohol, coffee, tea, and cola intake;
* inability to give written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with (a) history of SNAS (coexistence of typical cutaneous and gastrointestinal symptoms); (b) positive Ni-patch test; (c) clinical improvement of at least 70% from baseline after 4 weeks of low-Ni diet; (d) positivity of a double-blind placebo-controlled oral Ni challenge (DBPCO).
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Dietary assessment | At enrollment
  Dietary assessment includes questionnaire on 1) drinking alcohol, 2) particular diet (such as vegetarian, vegan or raw food), 3) number of meals per day, 4) same time for meals, 5) place of lunch on non-holiday, 6) frequency of eat away from home (times per week), 7) water intake, and 8) frequency of consumption of foods (desserts, processed meat, red meat, eggs, legumes, milk and derivatives, white meat, bread/pasta/rice, fish fruit and vegetable).
Change of body mass index (BMI) | Change from Baseline BMI at 15 and 30 days
  Collection of weight in kilograms and height in meters will be combined to report BMI in kg/m^2.
Change of circumference of wrist | Change from Baseline circumference of wrist at 15 and 30 days
  Collection of anthropometric data: circumference of wrist in centimeters.
Change of circumference of arm | Change from Baseline circumference of arm at 15 and 30 days
  Collection of anthropometric data: circumference of arm in centimeters.
Change of circumference of waist | Change from Baseline circumference of waist at 15 and 30 days
  Collection of anthropometric data: circumference of waist in centimeters.
Change of circumference of hip | Change from Baseline circumference of hip at 15 and 30 days
  Collection of anthropometric data: circumference of hip in centimeters.

SECONDARY OUTCOMES:
State of well-being | At enrollment, after 30 days
  Each patient answers SF-36v2 (Italian version) questionnaire. It comprises 36-items measuring eight dimensions of general QoL. Each question's score is coded, summed up, and transformed to a scale of 0 (worst possible health state measured by the questionnaire) to 100 (best possible health state).
Adherence to dietary therapy | After 15 days, after 30 days
  Assessment of adherence to dietary therapy through question "How many days a week did you adhere to the prescribed dietary treatment? - Two possible mutually exclusive answers: 1) <5 days a week, 2) ≥ 5 days a week.

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Nucera, Prof., MD, Principal Investigator — Università Cattolica del Sacro Cuore, Rome, Italy; Antonio Gasbarrini, Prof., MD, Study Director — Università Cattolica del Sacro Cuore, Rome, Italy
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No